CLINICAL TRIAL: NCT01586715
Title: A Phase IIa Clinical Trial to Study the Treatment of the Extremely Complex and Conventional Treatment Resistant Perianal Fistulae With Autologous Stem Cells From Lipoaspirate
Brief Title: Stem Cells Treatment for Extremely Complex Fistulae (HULPCIR)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HULPCIR-2010-01; 2010-024329-19 (EudraCT Number)
Record Dates: First submitted 2012-04-23; First posted 2012-04-27 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2012-04

CONDITIONS: Extremely Complex Perianal Fistulae
Keywords: Extremely complex perianal fistula; Adipose Derived Stem Cells

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Autologous Stem Cells (Experimental)
  Interventions: Drug: Adipose-derived stem cells without expanded

INTERVENTIONS:
Drug: Adipose-derived stem cells without expanded — Administration will be intralesional injection of cells suspension. They will be placed into fistula walls

SUMMARY:
The purpose of this study is to evaluate the practicability of the autologous e-ASC (Autologous Stem Cells) for the treatment of extremely complex and treatment resistant perianal fistulae.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Extremely Complex perianal fistulae
* Men and women over 18 years old. Good general state of health according to the findings of the clinical history and the physical examination
* Previous failure in at least one closing fistula standard treatment

Exclusion Criteria:

* Presence of severe proctitis or dominant active luminal disease requiring immediate therapy
* Patients with an abscess unless a complete toilet of the area with drainage of the collections and the absence of abscess and other collections is confirmed prior to treatment start
* Patients with a history of abuse of alcohol or other addictive substances in the 6 months prior to inclusion
* Patients with malignant tumor, except for basal cell or cutaneous squamous cell carcinoma, or patients with a prior history of malignant tumors, unless the neoplastic disease has been in remission for the previous 5 years
* Patients with cardiopulmonary disease which, in opinion of the investigator, in unstable or sufficiently serious to exclude the patient from the study.
* Patients with any type of medical or psychiatric disease which, in the opinion of the investigator, could be grounds for exclusion from study
* Patients with congenital or acquired immunodeficiencies. HIV, HBV, HCV or treponema infection, whether active or latent
* Patients who have suffering major surgery or severe trauma in the prior 6 months
* Pregnant or breastfeeding women
* Patients currently receiving, or having received within 1 month prior to enrollment into this clinical trial, any investigational drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2012-03; Primary Completion 2013-05 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Safety of treatment of extremely complex perianal fistulae. Percentage of treated extremely complex perianal fistulae and percentage of subjects with closed fistulae | 16 weeks
  Safety by control the adverse effects associated with treatment Fistula close by 3D ultrasound

SECONDARY OUTCOMES:
Quality of life assessment using the SF-12 Questionnaire | 1, 4, 16,24 weeks
  Test SF-12 of quality of life
Adverse events | 1, 4, 12, 24 weeks
  Control by investigation team of CRD (data collections)

CONTACTS AND LOCATIONS:
Overall Officials: Damián García Olmo, Prof MD, Principal Investigator — General Surgery Department (Hospital Universitario La Paz) and Cell Therapy laboratory
Locations (1):
- Hospital Universitario La Paz, Madrid, Madrid, Spain

REFERENCES:
- [Background] Bey NM. A new technique in dealing with superior rectovaginal fistulae. J. Obstrt Gynecol 1934. 41: 579-587
- [Background] Given FT Jr. Rectovaginal fistula. A review of 20 years' experience in a community hospital. Am J Obstet Gynecol. 1970 Sep 1;108(1):41-6. No abstract available. PMID 4916866
- [Background] Daniels BT. Rectovaginal fistula: a clinical and pathological study. Doctoral dissertation. Minneapolis: University of Minnesota 1949
- [Background] LAIRD DR. Procedures used in treatment of complicated fistulas. Am J Surg. 1948 Dec;76(6):701-8. doi: 10.1016/s0002-9610(48)90211-6. No abstract available. PMID 18895064
- [Background] Hoexter B, Labow SB, Moseson MD. Transanal rectovaginal fistula repair. Dis Colon Rectum. 1985 Aug;28(8):572-5. doi: 10.1007/BF02554145. PMID 4017820
- [Background] Fry RD, Shemesh EI, Kodner IJ, Timmcke A. Techniques and results in the management of anal and perianal Crohn's disease. Surg Gynecol Obstet. 1989 Jan;168(1):42-8. PMID 2909131
- [Background] Radcliffe AG, Ritchie JK, Hawley PR, Lennard-Jones JE, Northover JM. Anovaginal and rectovaginal fistulas in Crohn's disease. Dis Colon Rectum. 1988 Feb;31(2):94-9. doi: 10.1007/BF02562636. PMID 3338350
- [Background] Tuxen PA, Castro AF. Rectovaginal fistula in Crohn's disease. Dis Colon Rectum. 1979 Jan-Feb;22(1):58-62. doi: 10.1007/BF02586761. No abstract available. PMID 421652
- [Background] Hellers G, Bergstrand O, Ewerth S, Holmstrom B. Occurrence and outcome after primary treatment of anal fistulae in Crohn's disease. Gut. 1980 Jun;21(6):525-7. doi: 10.1136/gut.21.6.525. PMID 7429313
- [Background] Bandy LC, Addison A, Parker RT. Surgical management of rectovaginal fistulas in Crohn's disease. Am J Obstet Gynecol. 1983 Oct 15;147(4):359-63. doi: 10.1016/s0002-9378(16)32225-6. PMID 6624806
- [Background] Bauer JJ, Sher ME, Jaffin H, Present D, Gelerent I. Transvaginal approach for repair of rectovaginal fistulae complicating Crohn's disease. Ann Surg. 1991 Feb;213(2):151-8. doi: 10.1097/00000658-199102000-00010. PMID 1992942
- [Background] Tsang CB, Madoff RD, Wong WD, Rothenberger DA, Finne CO, Singer D, Lowry AC. Anal sphincter integrity and function influences outcome in rectovaginal fistula repair. Dis Colon Rectum. 1998 Sep;41(9):1141-6. doi: 10.1007/BF02239436. PMID 9749498
- [Background] Andreani SM, Dang HH, Grondona P, Khan AZ, Edwards DP. Rectovaginal fistula in Crohn's disease. Dis Colon Rectum. 2007 Dec;50(12):2215-22. doi: 10.1007/s10350-007-9057-7. Epub 2007 Sep 11. PMID 17846837
- [Background] García Olmo D, García-Verdugo JM, Alemany J, Gonzalez M, Gutierrez-Fuentes JA. CELL THERAPHY . Ed. Mac Graw Hill. Madrid 2007
- [Background] Aggarwal S, Pittenger MF. Human mesenchymal stem cells modulate allogeneic immune cell responses. Blood. 2005 Feb 15;105(4):1815-22. doi: 10.1182/blood-2004-04-1559. Epub 2004 Oct 19. PMID 15494428
- [Background] Puissant B, Barreau C, Bourin P, Clavel C, Corre J, Bousquet C, Taureau C, Cousin B, Abbal M, Laharrague P, Penicaud L, Casteilla L, Blancher A. Immunomodulatory effect of human adipose tissue-derived adult stem cells: comparison with bone marrow mesenchymal stem cells. Br J Haematol. 2005 Apr;129(1):118-29. doi: 10.1111/j.1365-2141.2005.05409.x. PMID 15801964
- [Background] Tse WT, Pendleton JD, Beyer WM, Egalka MC, Guinan EC. Suppression of allogeneic T-cell proliferation by human marrow stromal cells: implications in transplantation. Transplantation. 2003 Feb 15;75(3):389-97. doi: 10.1097/01.TP.0000045055.63901.A9. PMID 12589164
- [Background] Chamberlain G, Fox J, Ashton B, Middleton J. Concise review: mesenchymal stem cells: their phenotype, differentiation capacity, immunological features, and potential for homing. Stem Cells. 2007 Nov;25(11):2739-49. doi: 10.1634/stemcells.2007-0197. Epub 2007 Jul 26. PMID 17656645
- [Background] Le Blanc K, Ringden O. Immunobiology of human mesenchymal stem cells and future use in hematopoietic stem cell transplantation. Biol Blood Marrow Transplant. 2005 May;11(5):321-34. doi: 10.1016/j.bbmt.2005.01.005. PMID 15846285
- [Background] Maccario R, Podesta M, Moretta A, Cometa A, Comoli P, Montagna D, Daudt L, Ibatici A, Piaggio G, Pozzi S, Frassoni F, Locatelli F. Interaction of human mesenchymal stem cells with cells involved in alloantigen-specific immune response favors the differentiation of CD4+ T-cell subsets expressing a regulatory/suppressive phenotype. Haematologica. 2005 Apr;90(4):516-25. PMID 15820948
- [Background] Barrett AJ, Rezvani K, Solomon S, Dickinson AM, Wang XN, Stark G, Cullup H, Jarvis M, Middleton PG, Chao N. New developments in allotransplant immunology. Hematology Am Soc Hematol Educ Program. 2003:350-71. doi: 10.1182/asheducation-2003.1.350. PMID 14633790
- [Background] Garcia-Olmo D, Garcia-Arranz M, Garcia LG, Cuellar ES, Blanco IF, Prianes LA, Montes JA, Pinto FL, Marcos DH, Garcia-Sancho L. Autologous stem cell transplantation for treatment of rectovaginal fistula in perianal Crohn's disease: a new cell-based therapy. Int J Colorectal Dis. 2003 Sep;18(5):451-4. doi: 10.1007/s00384-003-0490-3. Epub 2003 May 20. PMID 12756590
- [Background] Garcia-Olmo D, Garcia-Arranz M, Herreros D, Pascual I, Peiro C, Rodriguez-Montes JA. A phase I clinical trial of the treatment of Crohn's fistula by adipose mesenchymal stem cell transplantation. Dis Colon Rectum. 2005 Jul;48(7):1416-23. doi: 10.1007/s10350-005-0052-6. PMID 15933795
- [Background] Garcia-Olmo D, Herreros D, Pascual I, Pascual JA, Del-Valle E, Zorrilla J, De-La-Quintana P, Garcia-Arranz M, Pascual M. Expanded adipose-derived stem cells for the treatment of complex perianal fistula: a phase II clinical trial. Dis Colon Rectum. 2009 Jan;52(1):79-86. doi: 10.1007/DCR.0b013e3181973487. PMID 19273960